CLINICAL TRIAL: NCT04879238
Title: Tailoring a Mindful Intervention to Enhance Opioid Treatment Outcomes in a Community Program
Brief Title: Tailoring a Mindful Intervention to Enhance Opioid Treatment
Acronym: BEING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Michael Fendrich, Associate Dean for Research, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20-0111
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Opioid-use Disorder
Keywords: Medication Assisted Treatment
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Yoga and Mindfulness intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga-Mindfulness Intervention (Experimental): Completing single session of yoga blended with mindfulness.
  Interventions: Behavioral: BEING

INTERVENTIONS:
Behavioral: BEING — 60 minute yoga session that blends mindfulness techniques
  Other Names: Yoga-Mindfulness

SUMMARY:
The main aim of this study is to better understand whether yoga can be blended with mindfulness as an additional intervention for people receiving medication assisted treatment at a Hartford-based community agency. If this program is acceptable to participants, then additional studies can allow us to determine its impact on stress and cravings. This intervention, developed by the researchers, is called BEING.

DETAILED DESCRIPTION:
This study is a micro-trial of our mindful yoga intervention, BEING, tailored to the MAT clients. This study adapts an existing manualized program of yoga and mindfulness intervention (BEING) for MAT participants. Particularly important is addressing potential challenges and concerns regarding acceptability and feasibility of implementation in vulnerable males with substance dependence. We are enlisting the support of a mindful yoga expert with experience in related populations (i.e., previously incarcerated male veterans with mental health issues) in the adaptation process. This study is designed primarily to test the feasibility of the implementation of the intervention. We cannot draw statistically valid conclusions about the impact the intervention on outcomes, given the overall study design. We plan to collect participant feedback on whether or not the intervention is acceptable. We also want to evaluate the availability, accessibility, acceptability and feasibility of collecting certain measures that would be collected in a subsequent adequately powered treatment study.

ELIGIBILITY:
Inclusion Criteria:

* Receiving Medication Assisted Treatment 18 years or older Released from incarceration within the past year Currently receiving services from the partnering community agency English speaking

Exclusion Criteria:

* Under 18 years old Non-English Speaking Current incarcerated Not receiving Medication Assisted Treatment Not receiving services from the partnering community agency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability | 3 months following pre-test
  Responses to questions about how acceptable participants found the intervention. The questions are indicated below: All questions can be responded to with one of the following answers:
  Completely disagree; disagree; neither agree nor disagree; agree; completely agree.
  I approve of the yoga and mindfulness training.
  I find the yoga and mindfulness training interesting.
  I like the yoga and mindfulness training.
  I welcome the yoga and mindfulness training.
  The training seems appropriate.
  The training applies to me.
  The training seems right for me.
  The training seems like a good match for me.
  The training seems easy to carry out.
  The training seems possible.
  The training seems doable.
  The training seems easy to use.
Adherence (self report) | 3 months following pre-test
  Adherence to MAT per client self report-Response to question on whether they are still on MAT.
Adherence (record review) | 3 months following intervention
  Review of client chart to see if the client is still on MAT and taking as prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fendrich, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Community Renewal Team, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Requests for participant data will be considered on an individual basis.